CLINICAL TRIAL: NCT04847661
Title: Efficacy of Mefloquine as Prophylaxis Against COVID-19: A Placebo-control, Randomized Clinical Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helwan University (Other)
Collaborators: Ain Shams University (Other); Fayoum University (Other); Assiut University (Other); Tanta University (Other); National Institute of Infectious Diseases, Tokyo, Japan (Unknown)
Responsible Party: Principal Investigator, Mohamed El Kassas, Associate professor and chief of Endemic Medicine Department, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 032
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Mefloquine

STUDY DESIGN:
Intervention Model Description: open-label, randomized, placebo controlled trial
Who Masked: Participant
Masking Description: The participants will be assigned randomly (locally in each center) in a 1:1 ratio to receive either Mefloquine (1100-1650 mg according to body weight), orally, or to receive the same number of placebo tablets (control group).Patients will be sequentially assigned a randomization number that was generated by an independent statistician. Randomization sequence will be provided in pre-sealed envelopes by the central co-ordination committee of the study. Individuals involved in randomization and masking will have no involvement in the rest of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mefloquine arm (Active Comparator): Mefloquine hydrochloride will be given in a dose of 1100-1650 mg, according to body weight (BW), splitted into two to three doses.
  * 30kg≤BW<45kg: 825mg followed by 275mg after 6-8 hours
  * 45kg≤BW<60kg: 825mg followed by 550mg after 6-8 hours
  * 60kg≤BW: 825mg followed by 550mg after 6-8 hours and then 275mg 6-8 hours after the second dose
  Interventions: Drug: Mefloquine as a prophylaxis against SARS-Cov-2 infection in household contacts of COVID 19 confirmed cases
- Control arm (Placebo Comparator): A similar tablet of non-active gradients was specifically manufactured for the study by EVA Pharma company. The placebo tablets exactly resemble the active treatment mefloquine tablets (the same shape, size and color).
  Interventions: Drug: Mefloquine as a prophylaxis against SARS-Cov-2 infection in household contacts of COVID 19 confirmed cases

INTERVENTIONS:
Drug: Mefloquine as a prophylaxis against SARS-Cov-2 infection in household contacts of COVID 19 confirmed cases — Mefloquine hydrochloride will be given in a dose of 1100-1650 mg, according to body weight (BW), splitted into two to three doses.

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Mefloquine as a prophylaxis against SARS-Cov-2 infection in household contacts of COVID 19 confirmed. This study is an open-label, randomized, placebo controlled trial.

A total of 1500 household contacts of COVID-19 confirmed cases who will attend triaging clinic of 5 Egyptian university centers (Helwan university hospital, Ain Shams university hospital, Assiut University Hospital, Fayoum university hospital and Tanta university hospital). The household contacts of COVID-19 confirmed subjects with a decision for home-isolation will be recruited to participate into this study. The recruited subjects from each center will be randomly assigned (locally in that center) into 2 groups (750 volunteer in each group). The 1st group will receive Mefloquine (1100-1650 mg according to body weight), orally, while the other group will receive the same number of placebo tablets (control group). Previous infection will be excluded for all recruited subjects by testing for the presence of anti-bodies against COVID-19 to exclude previous infection. Subjects who are tested negative will be allocated into one of the 2 study groups after randomization, and treatment will be started immediately (either mefloquine or placebo). In addition, a nasopharyngeal swap will be taken from each recruited subject and tested by PCR for COVID-19 to exclude current infection. After having the PCR results, positive cases will be analyzed separately to test for the disease severity.

Neurological and cardiac assessment will be done for all volunteers before recruitment to exclude the presence of any contraindication for Mefloquine intake. Both groups will be followed up clinically to detect any symptom or sign of COVID-19 infection for 2 weeks (during the period of home isolation). Nasopharyngeal swap with PCR for COVID-19 will be done for all included subjects at the end of the follow-up period (14 days), or at the appearance of symptoms or signs suggesting COVID-19 infection.

Primary end points of the study are either:

* End of follow up period (2 weeks)
* Confirmed diagnosis of COVID-19 infection during the study time Initial severity assessment of COVID-19 infection will be done in all infected subjects in both groups to compare severity, in addition to following up of the fate of the infected subjects.

DETAILED DESCRIPTION:
Aim:

To evaluate the efficacy and safety of Mefloquine as a prophylaxis against SARS-Cov-2 infection in household contacts of COVID 19 confirmed cases.

Primary objectives:

* Evaluating the role of Mefloquine in preventing SARS-Cov-2 infection
* Evaluation of the side effects that may result from the usage of Mefloquine.

Secondary objectives:

• Comparing the clinical severity/outcome of COVID-19 disease in infected subjects who received Mefloquine compared to those who did not receive the drug.

Patients and methods:

Study design:

This study is an open-label, randomized, placebo controlled trial. A total of 1500 household contacts of COVID-19 confirmed cases who will attend triaging clinic of 5 Egyptian university centers (Helwan university hospital, Ain Shams university hospital, Assiut University Hospital, Fayoum university hospital and Tanta university hospital). The household contacts of COVID-19 confirmed subjects with a decision for home-isolation will be recruited to participate into this study. The recruited subjects from each center will be randomly assigned (locally in that center) into 2 groups (750 volunteer in each group). The 1st group will receive Mefloquine (1100-1650 mg according to body weight), orally, while the other group will receive the same number of placebo tablets (control group). Previous infection will be excluded for all recruited subjects by testing for the presence of anti-bodies against COVID-19 to exclude previous infection. Subjects who are tested negative will be allocated into one of the 2 study groups after randomization, and treatment will be started immediately (either mefloquine or placebo). In addition, a nasopharyngeal swap will be taken from each recruited subject and tested by PCR for COVID-19 to exclude current infection. After having the PCR results, positive cases will be analyzed separately to test for the disease severity.

Neurological and cardiac assessment will be done for all volunteers before recruitment to exclude the presence of any contraindication for Mefloquine intake. Both groups will be followed up clinically to detect any symptom or sign of COVID-19 infection for 2 weeks (during the period of home isolation). Nasopharyngeal swap with PCR for COVID-19 will be done for all included subjects at the end of the follow-up period (14 days), or at the appearance of symptoms or signs suggesting COVID-19 infection.

Primary end points of the study are either:

* End of follow up period (2 weeks)
* Confirmed diagnosis of COVID-19 infection during the study time Initial severity assessment of COVID-19 infection will be done in all infected subjects in both groups to compare severity, in addition to following up of the fate of the infected subjects.

Written informed consent will be obtained from all participants. The trial will be conducted in accordance with the principles of the Declaration of Helsinki and the Good Clinical Practice guidelines of the International Conference on Harmonisation. The investigators vouch for data completeness and accuracy and adherence to the trial protocol.

Inclusion criteria:

This study will include volunteers household contact of COVID 19 confirmed cases who attend the triage clinic in the participating centers. Included persons should be > 18 years old and below 65 years, without any contraindications for Mefloquine usage.

Exclusion criteria:

* People with history of previous confirmed COVID-19 infection.
* Pregnant and lactating females.
* People with neuropsychiatric disorders: myasthenia gravis, epilepsy, psychotic disorder, schizophrenia, repeated episodes of anxiety, depression.
* People with liver cirrhosis or raised liver enzymes.
* People with arrhythmias or prolonged QT interval on EKG.
* People with a history of Quinidine-Quinine analogs allergy.

Mefloquine dose:

Mefloquine hydrochloride will be given in a dose of 1100-1650 mg, according to body weight (BW), splitted into two to three doses.

* 30kg≤BW<45kg: 825mg followed by 275mg after 6-8 hours
* 45kg≤BW<60kg: 825mg followed by 550mg after 6-8 hours
* 60kg≤BW: 825mg followed by 550mg after 6-8 hours and then 275mg 6-8 hours after the second dose Placebo A similar tablet of non-active gradients was specifically manufactured for the study by EVA Pharma company. The placebo tablets exactly resemble the active treatment mefloquine tablets (the same shape, size and color).

Blinding and randomization The participants will be assigned randomly (locally in each center) in a 1:1 ratio to receive either Mefloquine (1100-1650 mg according to body weight), orally, or to receive the same number of placebo tablets (control group).Patients will be sequentially assigned a randomization number that was generated by an independent statistician. Randomization sequence will be provided in pre-sealed envelopes by the central co-ordination committee of the study. Individuals involved in randomization and masking will have no involvement in the rest of the trial.

Data and Safety Monitoring Board (DSMB) DSMB will be appointed by the study principal investigator. The suggested committee will be independent from the investigator team. DSMB will be responsible for 1) periodically review and evaluate the accumulated study data for participant safety, study conduct and progress, and, when appropriate, efficacy, and 2) make recommendations to the investigator team concerning the continuation, modification, or termination of the trial.

Clinical and Laboratory Monitoring:

COVID-19 antibodies (rapid test; IgG and IgM) will be done before randomization; positive test result will be an exclusion critera, while those with negative results will be included in the study. Clinical, Laboratory data, and nasopharyngeal swab results will be done and recorded at the time of randomization and after 2 weeks, or when symptoms or signs of COVID-19 infection appeared.

Infection will be checked through quantitative real-time RT-PCR testing for serial oropharyngeal swab samples obtained at the same dates.

Outcome Measures:

1. Efficacy outcomes:

   1. The efficacy of Mefloquine will be measured by the detection of the difference in the rate of COVID-19 infection in both groups from the time of randomization.
   2. Severity of the disease for those infected during the study period.
2. Safety Outcomes:

Safety outcomes including adverse events that will occur during treatment, serious adverse events, and premature discontinuation of treatment will be assessed and classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

Egyptian team

1. Primary PI of the trial: Ass. Prof/ Mohamed El Kassas
2. Site PI for Helwan Univesity hospital: Ass. Prof/ Mohamed El Badry
3. Site PI for Ain Shams Univesity hospital: Prof/Hany Dabbous
4. Site PI for Tanta Univesity hospital: Prof/ Mohamed Samir
5. Site PI for Assiut Univesity hospital: Dr/Mohamed Ahmed Medhat
6. Site PI for Fayum Univesity hospital: Ass. Prof/Esam Ali Hassan
7. Data management: Prof. Sameera Ezzat, National Liver Institute, Menufia University
8. Clinical pharmacist in each center.
9. Clinical pathology specialist in each cener.
10. Data entery specialist Statistical Analysis Sample size: 1500 volanteer (750 in each group). We are planning a study of independent 2 groups with 1 control(s) per case. Prior data indicate that the incidence of infection among controls is 15%. If the true incidence of infection rate for experimental subjects is 10%, we will need to study 686 experimental subjects and 686 control subjects to be able to reject the null hypothesis that the failure rates for experimental and control subjects are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. Based on this calculation, a total of 750 subject in each group will be calculated to compensate for the droup outs.

Statistical methods The data will be analyzed by SPSS V. 23 (SPSS Inc. Released 2015. IBM SPSS statistics for windows, version 23.0, Armnok, NY: IBM Corp.). Data will be expressed in Number (No), percentage (%) mean (x̅), and standard deviation (SD). OneWay ANOVA is a test of significance that will be used for comparison of quantitative variables of normally distributed data. In contrast, the Kruskal-Wallis test will be used for the comparison of quantitative variables between three groups of not normally distributed data.

Primary efficacy analysis will be on an intention-to-treat basis and will include all the persons who will be randomized. The time to clinical improvement will be described by Kaplan-Meier plot and compared with a log-rank test. Hazard ratios with 95% confidence intervals will be calculated through the Cox proportional-hazards model.

Equipment All participating centers are well equipped with the necessary equipment; either for patients care, laboratory testing, or radiology services.

Cofedinitiality:

A. Protection of Subject Privacy - All volunteers are assured of their confidentiality both verbally and in the informed consent forms. The facilities are strictly limited to the staff of the research institution, clinics and to research volunteers. This is accomplished by a variety of stringent security measures. All medical records are to be stored in locked areas. Access to these areas is limited to the clinical support staff and the PI of the study. Volunteers' medical records are filed according to ID numbers. All forms on the chart, with the exception of consent form, display only the ID number.

B. Database Protection - Electronic data storage is similarly restricted with only the data management staff having access to databases containing confidential clinical records, i.e. those containing name or other identifying information.

C. Confidentiality during AE Reporting - Adverse events will be reported to the study PI, DSMB and notified to the IRB throughout the trial. Adverse event data will be analyzed quarterly, but serious or life-threatening adverse events require immediate reporting and follow-up. AE reports and quarterly summaries will not include subject-identifiable material. Each will include the identification code only.

Safety review plan and study termination The study PI will monitor the progress of the study weekly, including reasons for attrition and whether all participants met entry criteria. Further, progress and safety will be reviewed quarterly. These progress reports will include information on recruitment, retention/attrition, and AEs and will be provided to the DSMB quarterly. DSMB will also receive a yearly report that details data relevant to the possible early termination of the study. We plan an interim analysis for possible early trial termination for superiority or futility of the experimental therapy. The interim analysis will be performed by an independent statistician. The analysis will be performed on the primary endpoint when 50% (n=750) of patients have been randomized and have completed the 14 days follow-up with the second nasopharyngeal swap done.

ELIGIBILITY:
Inclusion Criteria:

* This study will include volunteers household contact of COVID 19 confirmed cases who attend the triage clinic in the participating centers. Included persons should be > 18 years old and below 65 years, without any contraindications for Mefloquine usage.

Exclusion Criteria:

* • People with history of previous confirmed COVID-19 infection.

  * Pregnant and lactating females.
  * People with neuropsychiatric disorders: myasthenia gravis, epilepsy, psychotic disorder, schizophrenia, repeated episodes of anxiety, depression.
  * People with liver cirrhosis or raised liver enzymes.
  * People with arrhythmias or prolonged QT interval on EKG.
  * People with a history of Quinidine-Quinine analogs allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The efficacy of Mefloquine | 2 weeks from randomization
  will be measured by the detection of the difference in the rate of COVID-19 infection in both groups from the time of randomization
Severity of COVID-19 | 2 weeks from randomization
  for those infected during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided